CLINICAL TRIAL: NCT04834583
Title: COVID-19 Pandemic and Small Businesses in the Health Care Sector - Work Environment, Health and Economy of Swedish Chiropractors and Naprapaths
Brief Title: Corona And Manual Professions
Acronym: CAMP
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Sophiahemmet University (Other)
Responsible Party: Principal Investigator, Iben Axen, Associate Professor, Karolinska Institutet
Other Study IDs: KIIMMRIAII
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will follow the chiropractors and naprapaths in Sweden to study how work environment, health, and economy is changing during the COVID-19 pandemic.

DETAILED DESCRIPTION:
All manual therapists that are members of a professional organization in Sweden will be invited to participate. The study started in November 2020 with follow-ups planned after 3,6 and 12 months.

All data-collection is taking place with digital questionnaires.

There are three main areas of interest:

1. Work environment (knowledge about viral contageon, protection, availability of protective measures, disturbances in care for patients)
2. Health (physical and psychological, how many caught the virus?)
3. Economy (income, costs, turnover)

ELIGIBILITY:
Inclusion Criteria:

* Chiropractor or naprapath working in Sweden
* clinically active
* belonging to a professional organization

Exclusion Criteria:

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Manual therapists, clinically active in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Work environment | 12 months
  Changes in routines according to the pandemic This includes systematic work environment routines, cleaning, wearing protective gear, not treating patients belonging to certain risk categories, changing appointment scheduling etc. There are no validated questionnaires to examine these concepts, as we have not experienced a pandemic in modern times, so the questions are constructed by the research group.
Physical Health -Pain | 12 months
  Physical pain using the Nordic Musculoskeletal Questionnaire
Psychological Health -depression | 12 months
  Depression assessed with DASS-21
Psychological Health -sleep | 12 months
  Sleep will be assessed using Karolinska Sleep Questionnaire.
Economy | 12 months
  Changes in company turnover. For clinic owners, this measure is assessing income and cost, estimated by clinic owners, There are no validated questionnaires to examine these concepts, as we have not experienced a pandemic in modern times, so the questions are constructed by the research group.

CONTACTS AND LOCATIONS:
Overall Officials: Iben Axén, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden